CLINICAL TRIAL: NCT05051137
Title: Comparison of Infliximab With Sulfasalazine/Hydroxychloroquine Initiated After Methotrexate by Rheumatoid Arthritis Patients Treated in Clinical Practice (Real-World Emulation of SWEFOT Trial)
Brief Title: Real-World Emulation of the SWEFOT Trial
Acronym: SWEFOT-RWEM
Status: Completed | Type: Observational
Sponsor: Karolinska Institutet (Other)
Collaborators: Harvard Medical School (HMS and HSDM) (Other)
Responsible Party: Principal Investigator, Thomas Frisell, Principal Investigator, Coordinator at the Clinical Epidemiology Division, Karolinska Institutet
Other Study IDs: SWEFOT-RWEM
Record Dates: First submitted 2021-09-10; First posted 2021-09-21 (Actual); Last update posted 2021-09-28 (Actual); Status verified 2021-09

CONDITIONS: Rheumatoid Arthritis
Keywords: Rheumatic Diseases
MeSH Terms: conditions — Arthritis, Rheumatoid; Rheumatic Diseases | interventions — Infliximab; CT-P13; Sulfasalazine; Hydroxychloroquine

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Infliximab initiators: Rheumatoid arthritis patients initiating infliximab after treatment with methotrexate for a minimum of 30 days.
  Interventions: Biological: Infliximab
- Sulfasalazine + Hydroxychloroquine initiators: Rheumatoid arthritis patients initiating sulfasalazine and hydroxychloroquine after treatment with methotrexate for a minimum of 30 days.
  Interventions: Drug: Sulfasalazine + Hydroxychloroquine

INTERVENTIONS:
Biological: Infliximab — Initiation of infliximab in any dose and frequency of administration. Could be discontinued for safety reasons and replaced by etanercept.
  Other Names: Flixabi, Inflectra, Remicade, Remsima, Zessly
  Groups: Infliximab initiators
Drug: Sulfasalazine + Hydroxychloroquine — Initiation of sulfasalazine and hydroxychloroquine not more than 180 days apart, in any dose and frequency of administration. Any one of the two drugs could be discontinued. while continuing the other, or both could be replaced by cyclosporine, for safety reasons.
  Other Names: Salazopyrin (sulfasalazine), Plaquenil (hydroxychloroquine)
  Groups: Sulfasalazine + Hydroxychloroquine initiators

SUMMARY:
This study will compare rheumatoid arthritis (RA) patients who have been treated in clinical practice with either infliximab or a combination of sulfasalazine and hydroxychloroquine, after having an active disease despite treatment with methotrexate for at least one month. To establish which patients respond to treatment, DAS28-ESR measurements (disease activity score using 28 joints and erythrocyte sedimentation rate) taken at treatment start and nine months thereafter, and the EULAR (European League Against Rheumatism) definition of a "good response" will be employed.

The purpose of the study is to verify if the same conclusion could be reached using data from patients treated in real world clinical practice as in a previous randomized controlled trial comparing the two treatment strategies (SWEFOT -- ClinicalTrials.gov Identifier: NCT00764725).

Inclusion criteria similar to the ones used in the emulated trial will be applied.

In real clinical practice, patients who receive infliximab may have more severe RA and may also differ in other ways from patients receiving sulfasalazine and hydroxychloroquine. To be able to compare the proportions of responders under each treatment in this "real-world" setting, the data will be re-weighted, so that patient characteristics become balanced between treatment groups.

DETAILED DESCRIPTION:
This observational study is designed to verify if the results of a previously conducted randomized controlled trial (SWEFOT -- ClinicalTrials.gov Identifier: NCT00764725) could be replicated with observational data, by emulating the trial protocol as close as possible.

Thus, early rheumatoid arthritis (RA) patients who initiated treatment with infliximab or a combination of sulfasalazine and hydroxychloroquine after at least 30 days of methotrexate will be identified in the Swedish Rheumatology Quality register (SRQ) linked to other Swedish national registers and will be compared. Similar inclusion/exclusion criteria to the ones used in SWEFOT will be applied. Also, in keeping with SWEFOT, the primary outcome is the proportion of patients with a "good EULAR response", measured nine months after study treatment initiation and considering patients who discontinued treatment before this point "non-responders" (i.e. "non-responder imputation" - regardless of the reason for discontinuation). For the combination of sulfasalazine and hydroxychloroquine the start of the second drug in the combination will be considered the study treatment initiation.

Since treatment assignment is not random in observational data, inverse probability of treatment weighting will be applied to balance patient characteristics between treatment cohorts, making them comparable (i.e. exchangeable). For each observation (i.e. patient), the probability of receiving the treatment actually received, conditional on a prespecified list of potential confounders will be estimated by logistic regression modelling and will be used to calculate a weight. Potential confounders included in the model are chosen based on knowledge about factors influencing treatment allocation and observed differences in such characteristics between treatment groups. The list of confounders includes: sex, age, country of origin, year of treatment start, duration of RA at treatment start, rheumatoid factor, disease activity at treatment start measured via: DAS28-ESR (disease activity score using 28 joints and erythrocyte sedimentation rate), CDAI (clinical disease activity index), number of swollen and tender joints, pain assessment (measured on a visual analogue scale) and HAQ-DI (health assessment questionnaire disability index), use of NSAIDs and of glucocorticoids, history of: cancer, diabetes, acute coronary syndrome, stroke, venous thromboembolism, peripheral vascular disease, obstructive respiratory disease, anaemia, psoriasis, neuropathies, pain, osteoporosis, depression or anxiety, joint surgery, retinopathy and hospitalized infections, the number of days spent in hospital within 5 years before treatment start, smoking status.

All data included in this study is extracted from Swedish national registers. In these registers, data is collected routinely, prospectively and independently from any study. Thus, data on baseline characteristics was collected before treatment initiation, while outcome data was recorded after treatment initiation.

The proportion of responders in each group and the ratio between proportions will be estimated using a weighted generalized linear model, specifying a binomial distribution for the dependent variable and a logarithmic identity function. Before analysis, missing data (covariates and outcome) will be imputed using fully conditional specification multiple imputation after non-responder imputation. All data-analysis (from weights estimation to responder-ratio estimation) will be conducted separately in each imputed data-set, the results being subsequently pooled using Rubin's rules.

ELIGIBILITY:
Inclusion criteria:

* Have started methotrexate less than 540 days after RA debut.
* Have used methotrexate for more then 30 days but less than 540 days before study treatment start.
* Have a baseline DAS28-ESR of more than 3.2 at study treatment start.
* Were residents of Sweden within 5 years before study treatment start

Exclusion criteria:

* Have used other DMARDs (antirheumatic drugs) than methotrexate before treatment start
* Have initiated study treatments later than May 2020

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients with rheumatoid arthritis as recorded in the Swedish Rheumatology Quality register (main data source), who initiated one of the two study treatments (infliximab or sulfasalazine + hydroxychloroquine). All eligible patients were included in the study (without any subsequent selection).
Sampling Method: Non-Probability Sample
Enrollment: 509 (Actual)
Dates: Start 2006-01-12 (Actual); Primary Completion 2020-11-16 (Actual); Study Completion 2020-11-16 (Actual)

PRIMARY OUTCOMES:
Good EULAR Response | 9 months after study treatment initiation
  The proportion of patients remaining on treatment and achieving a "good EULAR response" defined as a DAS28-ESR ≤ 3.2 at evaluation and a decrease > 1.2 units compared to the value at treatment initiation.

SECONDARY OUTCOMES:
Good or Moderate EULAR Response | 9 months after study treatment initiation
  The proportion of patients remaining on treatment and achieving a "good or moderate EULAR response" defined as a DAS28-ESR ≤ 5.1 at evaluation and a decrease > 0.6 units compared to the value at treatment initiation, or a DAS28-ESR > 5.1 at evaluation and a decrease > 1.2 units compared to treatment start.

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Frisell, PhD, Principal Investigator — Karolinska Institutet
Locations (1):
- Karolinska Institutet, Department of Medicine Solna, Clinical Epidemiology Unit, Stockholm, Sweden

IPD SHARING:
Plan to Share IPD: No
There is not a plan to make IPD available

REFERENCES:
- [Background] van Vollenhoven RF, Ernestam S, Geborek P, Petersson IF, Coster L, Waltbrand E, Zickert A, Theander J, Thorner A, Hellstrom H, Teleman A, Dackhammar C, Akre F, Forslind K, Ljung L, Oding R, Chatzidionysiou A, Wornert M, Bratt J. Addition of infliximab compared with addition of sulfasalazine and hydroxychloroquine to methotrexate in patients with early rheumatoid arthritis (Swefot trial): 1-year results of a randomised trial. Lancet. 2009 Aug 8;374(9688):459-66. doi: 10.1016/S0140-6736(09)60944-2. PMID 19665644
- [Background] van Vollenhoven RF, Geborek P, Forslind K, Albertsson K, Ernestam S, Petersson IF, Chatzidionysiou K, Bratt J; Swefot study group. Conventional combination treatment versus biological treatment in methotrexate-refractory early rheumatoid arthritis: 2 year follow-up of the randomised, non-blinded, parallel-group Swefot trial. Lancet. 2012 May 5;379(9827):1712-20. doi: 10.1016/S0140-6736(12)60027-0. Epub 2012 Mar 29. PMID 22464340